CLINICAL TRIAL: NCT04262960
Title: Effect of Continuous Positive Airway Pressure on Chronotype, Dietary Intake, and Cardiovascular Risk Markers of Elderly Patients With Obstructive Sleep Apnea
Brief Title: Effect of Continuous Positive Airway Pressure on Chronotype, Dietary Intake, and Cardiovascular Risk Markers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 07034918000005327
Record Dates: First submitted 2020-01-15; First posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Obstructive Sleep Apnea of Adult
Keywords: Obstructive sleep apnea; Continuous positive airway pressure; Elders; Chronotype; Cardiovascular risk; Food intake
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active CPAP (Active Comparator): auto-PAP with therapeutic pressure
  Interventions: Device: Device: active CPAP
- sham-CPAP (Sham Comparator): auto-PAP with pressure less than 1cm H2O
  Interventions: Device: Device: sham-CPAP

INTERVENTIONS:
Device: Device: active CPAP — auto-PAP with pressure between 4 and 20 cm H2O will be administered to randomized patients
  Arms: active CPAP
Device: Device: sham-CPAP — The sham-CPAP will be fixed in the lowest pressure (4cmH2) and modified as recommended by Farré et al, with pressure that no greater than 1cm H2O.
  Arms: sham-CPAP

SUMMARY:
In this study the investigators will evaluate chronotype, food intake pattern, and cardiovascular risk markers of elder individuals with OSA, in use of CPAP, when submitted to two weeks of CPAP withdrawal.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a growing public health problem affecting up to 95% of older populations. This sleep disorder influences glucose metabolism, leptin and grelin levels, promotes sympathetic overactivity, and is associated to increased cardiovascular events. All awake-sleep processes are determined by clock-genes and by external factors such as sunlight, physical activity, feeding, sleep, and chronotype. Chronotype is the propensity for the individual to wake and sleep at a particular time during a 24-hour period, and is categorized as morning, intermediate or evening chronotype. Individuals with morning chronotype are more alert in the morning and choose an earlier bedtime. Individuals with evening chronotype have more inclination for evening activities and choose a later bedtime. And those classified as intermediate chronotype show low or no preference for either morning or evening hours for activities. Individuals with evening chronotype tend to have higher nocturnal food intake, body mass index (BMI), levels of stress hormones, and more sleep apnea episodes. In humans, changes in sleep pattern for a few days are sufficient to affect food intake pattern. Two days of partial sleep deprivation increases hunger and appetite for calorie-dense foods with high carbohydrate content. Food composition, quantity, timing, and rhythmicity of meals impact on microbiota and metabolism, increasing basal level of inflammation and age related diseases. The aging process comes with an increase in the molecules involved in hypercoagulable states, such as plasminogen activator inhibitor 1 (PAI-1), a protein induced by inflammatory mediators, which creates a prothrombotic state, resulting in a pathological deposit of fibrin followed by tissue damage. The increase in PAI-1 expression is related to the development of tissue pathologies such as thrombosis, fibrosis and cardiovascular disease. Adults with moderate-to-severe OSA have higher levels of PAI-1, and respond to two weeks of Continuous Positive Airway Pressure (CPAP) with a 50% reduction in this antifibrinolytic enzyme. The impact of CPAP use on chronotype, food intake pattern, and cardiovascular risk markers have never been studied in elder individuals with OSA.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 to 75 years
* Previous diagnosis of OSA with AHI> 30 events / hour
* Body mass index below 34,9 kg/m2
* Use of CPAP for more than one year, with an average duration of at least 6 hours per night, confirmed by the device's memory
* Evidence in the device that you have stopped using it previously, for at least two weeks, with no relevant symptoms
* Use of automatic CPAP device with full memory for at least one year, preferably using device model with internet data access
* Subjects physically active and willing to provide informed consent
* Subjects willing to attend visits and blood collections in series

Exclusion Criteria:

* History of myocardial infarction, stroke or transient ischemic attack (TIA) or peripheral vascular disease.
* History of chronic diseases such as diabetes mellitus ( A fasting plasma glucose (FPG) level of 152 mg/dL or A1C > 7,5 % ), uncontrolled severe hypertension (SBP >180 DBP > 110), renal failure on dialysis, cancer, autoimmune or liver disease
* A significant history of medical or psychiatric disease that may decompensate with altered sleep patterns or impair participation in the trial
* Severe or unstable clinical conditions that may be exacerbated by discontinuation of CPAP (cardiac, pulmonary, renal or other organ disorders not yet treated or worsening of symptoms in the last two months, eg cardiac arrhythmias, congestive heart failure and oxygen-dependent lung disease)
* Another primary sleep disorder that requires intervention with medications.
* Patients with unusual sleep or wake habits, including shift work.
* Professional driver or who crosses paths of more than one hour driving, in which the s sleepiness can be risk of accident.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
The association between withdrawal CPAP with chronotype, food intake pattern and cardiovascular risk markers. | 4 weeks
  Chronotype as defined by the MEQ chronotype categories; food intake pattern dietary assessed by a 3 day food intake diary, and Plasminogen activator inhibitor type 1 (pg/mL) and plasminogen (ng/mL) measured from blood samples by ELISA.

SECONDARY OUTCOMES:
Plasminogen activator inhibitor type 1 | 1 week before and two weeks after randomization
  Plasminogen activator inhibitor type 1 (pg/mL) measured from a blood sample by ELISA.
Plasminogen | 1 week before and two weeks after randomization
  Plasminogen (ng/mL) measured from a blood sample by ELISA.
Blood pressure | 1 week before and two weeks after randomization
  We will be measuring Systolic and Diastolic Blood Pressure by Ambulatory 24-hour blood pressure monitoring.
Chronotype | 1 week before and 1 week after randomization - MEQ 1 week before and 2 weeks after randomization
  Morningness Eveningness Questionaire (MEQ) inquires about daily performance and preferred sleep schedule (score range 16 to 86) and presents 19 questions. Based on their scores, individuals will be classified as morning (score: 50-86) or evening type (score: 16-49).
Sleep habits | 1 week before and 1 week after randomization - MEQ 1 week before and 2 weeks after randomization
  Sleeping and awake periods will be assessed by a wrist actigraphy monitor (ActTrust, Condor Instruments, São Paulo - Brazil) according to the Cole-Kripke algorithm, and the duration expressed in minutes.
Dietary intake | For three days before and after randomization
  Participants will record food intake for three consecutive days, including two days of the week and one day of the weekend. During the visit, they will receive verbal instructions on how to register, as well as written instructions consisting of printed material showing the portion sizes of the food and how to fill the journal. Information about mealtimes will also be obtained. Data will be analyzed using a Brazilian Nutrition Software (Dietbox) and expressed in calories an in percentage of total caloric intake. A meal will be considered as an occasion to eat when consumption exceeds 20 kcal. Higher caloric intake in the evening will be associated to evening chronotype.
Autonomic modulation | 1 week before and two weeks after randomization
  Autonomic modulation will be evaluated by low frequency (LF) and high frequency (HF) components of heart rate spectral analysis, at rest and during sympathetic stimulation with the Stroop Color Word Test, expressed in ms2/Hz and in normalized units. The amount of increase in LF/HF ratio during sympathetic stimulation will reflect the autonomic modulation integrity.

CONTACTS AND LOCATIONS:
Overall Officials: Ruy Silveira Morais Filho, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No